CLINICAL TRIAL: NCT05239052
Title: The Feasibility and Effect of Physical Activity With Computerized Upper Limb Training Strategy on Health Promotion for Stroke Wheelchair User in Long-term Care Institution
Brief Title: The Feasibility and Effect of PACUTS on Health Promotion for Stroke Wheelchair User in Long-term Care Institution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20180035
Record Dates: First submitted 2022-01-06; First posted 2022-02-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2018-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer intervention group (Experimental): stroke subjects with wheelchair users completed computer screen tasks with affected arm or bilateral arm movement
  Interventions: Other: computer task intervention
- conventional long-term care services group (Active Comparator): stroke subjects with wheelchair users receive conventional long-term care services
  Interventions: Other: conventional long-term care services

INTERVENTIONS:
Other: computer task intervention — subject received programs for upper arm movement training with providing computer screen task activities
  Arms: computer intervention group
Other: conventional long-term care services — stroke subjects with wheelchair users receive conventional long-term care services
  Arms: conventional long-term care services group

SUMMARY:
Most of the residents in long-term care institution were wheelchair users, however, it would limit the participation in physical activities, and thus increase the degree of disability as they excessively rely on wheelchair. Recently, with the development of rehabilitation technology, the clients can receive more individualized physical activities intervention. Moreover, using technology as an assistive modality would reduce the demand of manpower, and provide higher treatment intensity with repeated training and objective performance feedback. Based upon our previous study finding from the physical activity with computerized upper limb training system (PACUTS), we propose to build a training strategy of physical activity for stroke wheelchair user in long-term care institution and to analyze its feasibility as well as the treatment effects, in the next two years.

The mixed method design will be applied. In the qualitative research, we will focus on the experience of physical activity training and subject's "adoption and acceptance" of the PACUTS. In terms of the quantitative research, 50 residents who currently live in long-term care institution will be recruited. Double-blinded randomized control-group pretest-posttest design will be conducted. In the experiment group, the participant will receive the intervention of PACUTS for 12 weeks/ 5 sessions per week/ 30 minutes, at least, per session. In terms of control group, the participant will receive a regular treatment program and physical activities scheduled by occupational therapist. This study is expected to contribute to build a training strategy with computerized upper limb training system which can helpfully promote the participation in physical activities and health outcomes for w/c residents living in long-term care institution.

DETAILED DESCRIPTION:
In the past few years, the government has been focusing on community based care, the idea so-called aging-in-place. Therefore, the intervention model for residents in long-term care institution had been noticed by the researcher. Most of the residents in long-term care institution were wheelchair users, however, it would limit the participation in physical activities, and thus increase the degree of disability as they excessively rely on wheelchair. Recently, with the development of rehabilitation technology, the clients can receive more individualized physical activities intervention. Moreover, using technology as an assistive modality would reduce the demand of manpower, and provide higher treatment intensity with repeated training and objective performance feedback. Based upon our previous study finding from the physical activity with computerized upper limb training system (PACUTS), we propose to build a training strategy of physical activity for stroke wheelchair user in long-term care institution and to analyze its feasibility as well as the treatment effects, in the next two years.

The mixed method design will be applied. In the qualitative research, we will focus on the experience of physical activity training and subject's "adoption and acceptance" of the PACUTS. Through in-depth interview, field notes and different interviewers, the qualitative data analysis with phenomenology design will be applied. In terms of the quantitative research, 50 residents who currently live in long-term care institution will be recruited. Double-blinded randomized control-group pretest-posttest design will be conducted. In the experiment group, the participant will receive the intervention of PACUTS for 12 weeks/ 5 sessions per week/ 30 minutes, at least, per session. In terms of control group, the participant will receive a regular treatment program and physical activities scheduled by occupational therapist. Participants will be assessed by outcome measures, including Time Up and Go Test, Box and Block Test, Grip Strength Assessment, the Ruff 2 & 7 Selective Attention Test, System Usability Scale, Barthel Index, SF-36 and the Falls Efficacy Scale-International. Descriptive statistics, independent-sample t test, paired-sample t test or mixed type 2-way ANOVA will be performed for data analysis. This study is expected to contribute to build a training strategy with computerized upper limb training system which can helpfully promote the participation in physical activities and health outcomes for w/c residents living in long-term care institution.

ELIGIBILITY:
Inclusion Criteria:

* Currently living in a long-term care institution
* Stoke, onset over 6 months
* Wheelchair user
* Maintain sitting 30 minutes
* No cognition impairment

Exclusion Criteria:

* Aphsia
* Dementia, Cancer and MS
* PNS impairment
* Cardiopulmonary dysfunction
* Visual impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Box and Block Test | pre-test, post-test(Change from pre-test Box and Block Test after 6 weeks' intervention)
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke.
Grip Strength Assessment | pre-test, post-test(Change from pre-test Grip Strength Assessment after 6 weeks' intervention)
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength.
System Usability Scale | only post-test(after 6 weeks' intervention)
  The System Usability Scale, or SUS, is a simple survey that provides a high-level score for the usability of a product.
Moss Attention Rating Scale | pre-test, post-test(Change from pre-test Moss Attention Rating Scale after 6 weeks' intervention)
  The MARS was designed as an observational rating scale to provide a reliable, quantitative and ecologically valid measure of attention-related behavior after TBI.
upper limb endurance | pre-test, post-test(Change from pre-test upper limb endurance after 6 weeks' intervention)
  can raise your hands several times in a minute

SECONDARY OUTCOMES:
Barthel Index | pre-test and post-test(after 6 weeks' intervention)
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.
The 12-Item Short Form Health Survey | pre-test and post-test(after 6 weeks' intervention)
  The 12-item Short Form Health Survey (SF-12) as a shorter alternative of the SF-36 is largely used in health outcomes surveys.
Falls Efficacy Scale-International | pre-test and post-test(after 6 weeks' intervention)
  are measures of "fear of falling" or, more properly, "concerns about falling", which are suitable for use in research and clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Jong Chang, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Department of Occupational Therapy, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: starting one year after publication
Access Criteria: For Meta-analysis study

REFERENCES:
- [Result] Chen KM, Li CH, Huang HT, Cheng YY. Feasible modalities and long-term effects of elastic band exercises in nursing home older adults in wheelchairs: A cluster randomized controlled trial. Int J Nurs Stud. 2016 Mar;55:4-14. doi: 10.1016/j.ijnurstu.2015.11.004. Epub 2015 Nov 28. PMID 26655368
- See also: Feasible modalities and long-term effects of elastic band exercises in nursing home older adults in wheelchairs: A cluster randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/26655368/